CLINICAL TRIAL: NCT00502840
Title: An Open Label Study to Evaluate the Safety of Re-treatment With MabThera, and Its Effect on Treatment Response, in Patients With Rheumatoid Arthritis Following Inadequate Response to a Single Anti-TNF Agent (Extension Study to ML19070).
Brief Title: A Study of Re-Treatment With MabThera (Rituximab) in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to a Single Anti-TNF Inhibitor.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19071
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1g iv on days 1 and 15

SUMMARY:
This single arm study will evaluate the efficacy and safety of repeated courses of MabThera in patients with active rheumatoid arthritis who have participated in ML19070, and have completed the week 24 visit. Eligible patients (DAS28 >2.6 after week 24), will receive 2 infusions of 1g MabThera (Day 1 and day 15). For all patients in this extension study, up to 3 repeated courses of treatment are allowed. The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with rheumatoid arthritis who participated in ML19070, and have completed the week 24 visit;
* eligible for re-treatment (DAS28 >2.6 after week 24, swollen joint count >=4, tender joint count >=4).

Exclusion Criteria:

* patients who have withdrawn from treatment in ML19070 pre-week 16;
* patients with a previous response in DAS28 <0.6 to MabThera after week 16;
* concurrent treatment with any DMARD except for methotrexate, any TNF alpha inhibitor, or other biologic or investigational agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2007-07-23 (Actual); Primary Completion 2011-09-20 (Actual); Study Completion 2011-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- Germany (51):
  - Rheumapraxis - Dres. Edmund Edelmann, Gerhard Straeßner und Hans Bloching, Bad Aibling
  - Rheuma-Klinikum Bad Bramstedt Klinik fuer Rheumatologie und Immunologie, Bad Bramstedt
  - Campus Charité Mitte Charité Centrum 12. Med.Klinik Abt.Rheumatologie u.Klin.Immunologie, Berlin
  - Praxis Dr. Silke Zinke, Berlin
  - Immanuel-Krankenhaus; Rheumklinik Berlin Buch, Berlin
  - Ev. Waldkrankenhaus Spandau; Klinik für Innere Medizin, Berlin
  - Ambulantes Rheumazentrum Dr.med. Helmut Sörensen, Berlin
  - Universitätsklinikum Bonn Med. Klinik u.Poliklinik III, Bonn
  - Klinik der Uni zu Köln; Klinik für Innere Medizin, Cologne
  - HELIOS Seehospital Sahlenburg Abt.Internist.Rheumatologie, Cuxhaven
  - Praxis PD Dr. med. Ekkehard Röther, Donaueschingen
  - Rheumatologisches MVZ Dresden GmbH, Dres. Holger Schwenke, Reiner Schwenke, Annekatrin Georgi, Dresden
  - Med. Versorgungszentrum Kästner + Kästner GbR Ambulantes Rheumazentrum, Erfurt
  - Universitätsklinikum Erlangen; Medizinische Klinik 3; Rheumatologie und Immunologie, Erlangen
  - Kliniken Essen; Süd Kath.Krankenhaus St.Josef; Abt. Rheumatologie und Immunologie, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Medizinische Klinik II; Abt. Rheumatologie, Frankfurt am Main
  - Universitätsklinikum Freiburg; Medizinische UNI-Klinik; Abt. Innere Medizin - VI Rheumatologie, Freiburg im Breisgau
  - Herz-Jesu-Krankenhaus Abt.Geriatrie u. Rheumatologie, Fulda
  - Universitätsklinikum Gießen und Marburg GmbH Standort Gießen Medizinische Klinik III, Giessen
  - MEDIGREIF Fachkrankenhaus fuer Rheumatologie und Orthopädie; Vogelsang-Gommern, Gommern
  - Evangelisches Krankenhaus Hagen-Haspe Rheumaklinik, Hagen
  - Universitätsklinikum Halle Klinik u.Poliklinik f.Innere Medizin I, Halle
  - Schön Klinik Hamburg-Eilbek Klinik für Rheumatologie, Hamburg
  - Medizinische Hochschule Zentrum Innere Medizin Abt.Klinische Immunologie und Rheumatologie, Hanover
  - Rheumapraxis PD Dr.med. Bernhard Heilig, Heidelberg
  - UNI-Klinikum Heidelberg Medizinische Klinik Innere Medizin V, Heidelberg
  - Rheumazentrum-Ruhrgebiet, St. Josefs-Krankenhaus; Rheumatologie, Herne
  - Universitaetsklinikum des Saarlandes; medizinische Klinik und Poliklinik; Innere Medizin I, Homburg/Saar
  - Universitätsklinikum Jena; Klinik für Innere Medizin III, Jena
  - Praxis Dr.med. Ursula Mauß-Etzler, Karlsruhe
  - Klinikum der Stadt Ludwigshafen; Medizinische Klinik A, Ludwigshafen
  - Praxis Andreas Reck, Mittelherwigsdorf
  - LMU München, Bereich Pettenkoferstr., Medizinische Poliklinik, München
  - Praxis Prof. Dr.med. Herbert Kellner, München
  - Gemeinschaftspraxis Prof. Dr. med. Klaus Krueger, Guenter Kellerer und Paul Kellerer, München
  - Universitätsklinikum Münster Innere Medizin B, Münster
  - Praxis Dr.med. Sylvia Berger, Naunhof
  - Evang.Krankenhaus Medizinische Klinik, Oldenburg
  - Rheumapraxis an der Hase, Osnabrück
  - Praxis Dr.med. Anett Gräßler, Pirna
  - Evangelisches Fachkrankenhaus; Rheumaklinik, Ratingen
  - Klinikum der Uni Regensburg; Klinik f.Innere Medizin I Abt. Hämatologie und Internistische Onkologie, Regensburg
  - Praxis Dr.med. Matthias Richter, Rostock
  - St.-Josef-Stift Klinik für Rheumatologie, Sendenhorst
  - Rheumatologische Schwerpunktpraxis am Feuersee, Stuttgart
  - Johanniter-Krankenhaus im Fläming Treuenbrietzen GmbH; Fachklinik Pneumologie/ Thoraxchirurgie, Treuenbrietzen
  - Universitätsklinikum Tübingen Medizinische UNI-Klinik und Poliklinik Abt. Innere Medizin II, Tübingen
  - Universitätsklinikum Ulm; Medizinische Uni-Klinik III Abt. Innere Medizin III Hämatologie u. Onkolo., Ulm
  - Praxis Dr.med. Wolf-Dieter Wörth, Wiesbaden
  - Medizinisches Zentrum Betriebsteil Marienhöhe Klinik f.Internistische Rheumatologie, Würselen
  - Universitätsklinikum Würzburg; Medizinische Klinik und Poliklinik II; Hämatologie / Onkologie, Würzburg

REFERENCES:
- [Derived] Dimanche A, Bervini D, Miller DR, Schar A, Goldberg J, Raabe A, Dunn AK. Cortical perfusion measurements with laser speckle contrast imaging during adenosine induced cardiac arrest for aneurysm clipping: a case report. Acta Neurochir (Wien). 2024 Jan 23;166(1):27. doi: 10.1007/s00701-024-05925-2. PMID 38261093

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Plus Methotrexate (MTX): Participants received rituximab 1 gram (g), intravenously (IV), and methylprednisolone 100 mg, IV, on Days 1 and 15 (one cycle). Participants should have been receiving mandatory background therapy with MTX (prescribed as necessary by the treating physician) at a stable dose between 7.5 and 25 milligrams (mg) weekly; participants may also have been receiving a stable dose of folic acid. Participants with Disease Activity Score Based on 28 Joint Count (DAS28) greater than or equal to (≥)2.6 and an improvement in DAS28 greater than (>0.6) 16 to 24 weeks following treatment could have received up to two additional cycles of rituximab treatment.
Period: Overall Study
Arm/Group | Rituximab Plus Methotrexate (MTX)
Started | 193
Completed | 93
Not Completed | 100
Not completed — Adverse Event | 5
Not completed — Additional or changed therapy | 48
Not completed — Lack of Efficacy | 11
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 6
Not completed — Administrative problems | 1
Not completed — Other | 20

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of the trial medication and had at least 1 safety follow-up, whether withdrawn prematurely or not. A safety follow-up was assumed if the participant had at least 1 documented study visit after baseline or if at least 1 adverse event had been documented with start date after baseline.
Groups:
- Rituximab Plus MTX: Participants received rituximab 1 g, IV, and methylprednisolone 100 mg, IV, on Days 1 and 15 (one cycle). Participants should have been receiving mandatory background therapy with MTX (prescribed as necessary by the treating physician) at a stable dose between 7.5 and 25 mg weekly; participants may also have been receiving a stable dose of folic acid. Participants with DAS28 ≥2.6 and an improvement in DAS28 >0.6 16 to 24 weeks following treatment could have received up to two additional cycles of rituximab treatment.
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 193
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DAS28 Score at Week 24
Description: DAS28 calculated from the swollen joint count (SJC) and tender joint count (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and Patient Global Asessment of disease activity (participant- rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). A clinically meaningful improvement in DAS28 was defined as an improvement of 1.2 units.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) Population: all participants who signed the informed consent form, received at least 1 dose of study medication, and where the DAS28 was measured at least once under study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Rituximab Plus MTX: Participants received rituximab 1 g, IV, and methylprednisolone 100 mg, IV, on Days 1 and 15 (one course of treatment). Participants should have been receiving mandatory background therapy with MTX (prescribed as necessary by the treating physician) at a stable dose between 7.5 and 25 mg weekly; participants may also have been receiving a stable dose of folic acid. Participants with DAS28 ≥2.6 and an improvement in DAS28 >0.6 16 to 24 weeks following treatment could have received up to two additional courses of rituximab treatment.
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale | -2.12 (1.41)

2. Secondary Outcome: DAS28 Score by Treatment Course and Follow-up (FU) Visit
Description: DAS28 was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The DAS28 consists of SJC and TJC measurements, the ESR (measured in mm/hr), and Patient Global Asessment of disease activity (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 less than or equal to (≤)3.2 equals (=) low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n (number) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=173) | 5.15 (1.09)
  Course 1: FU Week 8 (n=171) | 4.09 (1.22)
  Course 1: FU Week 16 (n=167) | 3.72 (1.29)
  Course 1: FU Week 24 (n=163) | 3.78 (1.25)
  Course 1: FU Month 9 (n=76) | 3.94 (1.56)
  Course 1: FU Month 12 (n=38) | 3.79 (1.38)
  Course 2: FU Week 8 (n=104) | 3.69 (1.25)
  Course 2: FU Week 16 (n=106) | 3.34 (1.04)
  Course 2: FU Week 24 (n=107) | 3.56 (1.26)
  Course 2: FU Month 9 (n=65) | 3.53 (1.34)
  Course 2: FU Month 12 (n=47) | 3.98 (1.50)
  Course 3: FU Week 8 (n=35) | 3.59 (1.09)
  Course 3: FU Week 16 (n=37) | 3.25 (1.07)
  Course 3: FU Week 24 (n=38) | 3.65 (1.39)
  Course 3: FU Month 9 (n=24) | 3.94 (1.33)
  Course 3: FU Month 12 (n=18) | 4.12 (1.22)

3. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response of 'Good' or 'Moderate' by Treatment Course
Description: DAS28 was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders had a change from baseline >1.2 with a DAS28 score ≤3.2; moderate responders had a change from baseline >1.2 with a DAS28 score >3.2 to ≤5.1 or a change from baseline >0.6 to ≤1.2 with a DAS28 score ≤5.1.
Time Frame: Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
percentage of participants
  Course 1 (n=173) | 78.0
  Course 2 (n=107) | 86.9
  Course 3 (n=38) | 86.8

4. Secondary Outcome: Percentage of Participants Achieving a Response By EULAR Category and Treatment Course
Description: Response was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders had a change from baseline >1.2 with a DAS28 score ≤3.2; moderate responders had a change from baseline >1.2 with a DAS28 score >3.2 to ≤5.1 or a change from baseline >0.6 to ≤1.2 with a DAS28 score ≤5.1; non-responders had a change from baseline ≤0.6 or change from baseline >0.6 and ≤1.2 with a DAS28 score > 5.1.
Time Frame: Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Groups:
- Rituximab Pluse MTX: Participants received rituximab 1 g, IV, and methylprednisolone 100 mg, IV, on Days 1 and 15 (one course of treatment). Participants should have been receiving mandatory background therapy with MTX (prescribed as necessary by the treating physician) at a stable dose between 7.5 and 25 mg weekly; participants may also have been receiving a stable dose of folic acid. Participants with DAS28 ≥2.6 and an improvement in DAS28 >0.6 16 to 24 weeks following treatment could have received up to two additional courses of rituximab treatment.
Arm/Group | Rituximab Pluse MTX
Number analyzed (Participants) | 173
percentage of participants
  Course 1: Good response (n=173) | 32.4
  Course 1: Moderate response (n=173) | 45.7
  Course 2: Good response (n=107) | 43.0
  Course 2: Moderate response (n=107) | 43.9
  Course 3: Good response (n=38) | 44.7
  Course 3: Moderate response (n=38) | 42.1

5. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Score by Treatment Course
Description: HAQ-DI was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The HAQ-DI score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. For each of the categories, participants reported the amount of difficulty they had in performing 2 or 3 specific sub-category items. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. The standard disability score was calculated from the 8 categories by dividing the sum of the individual categories by the number of categories answered ;total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. The questionnaire was provided in a German translation and was scored based on the instructions from the Stanford University Medical Center.
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=173) | 1.43 (0.64)
  Course 1: FU Week 8 (n=171) | 1.36 (0.68)
  Course 1: FU Week 16 (n=164) | 1.31 (0.67)
  Course 1: FU Week 24 (n=164) | 1.28 (0.68)
  Course 1: FU Month 9 (n=76) | 1.33 (0.72)
  Course 1: FU Month 12 (n=39) | 1.29 (0.84)
  Course 2: FU Week 8 (n=100) | 1.31 (0.62)
  Course 2: FU Week 16 (n=104) | 1.26 (0.61)
  Course 2: FU Week 24 (n=106) | 1.22 (0.59)
  Course 2: FU Month 9 (n=65) | 1.34 (0.62)
  Course 2: FU Month 12 (n=49) | 1.38 (0.65)
  Course 3: FU Week 8 (n=34) | 1.25 (0.63)
  Course 3: FU Week 16 (n=37) | 1.25 (0.67)
  Course 3: FU Week 24 (n=38) | 1.25 (0.63)
  Course 3: FU Month 9 (n=25) | 1.12 (0.59)
  Course 3: FU Month 12 (n=17) | 1.35 (0.57)

6. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score by Treatment Course
Description: FACIT-F was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The FACIT fatigue scale is based on a 13-item questionnaire to assess the therapy-induced fatigue. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (best) to 52 (worst). The assessment was originally developed for chronic illnesses and is now validated for patients with rheumatoid arthritis (RA). The questionnaire was provided in a German translation.
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=169) | 20.16 (11.37)
  Course 1: FU Week 8 (n=165) | 18.48 (11.39)
  Course 1: FU Week 16 (n=157) | 18.81 (12.14)
  Course 1: FU Week 24 (n=161) | 17.75 (11.76)
  Course 1: FU Month 9 (n=72) | 18.17 (12.53)
  Course 1: FU Month 12 (n=35) | 20.77 (13.48)
  Course 2: FU Week 8 (n=99) | 16.43 (11.18)
  Course 2: FU Week 16 (n=101) | 16.19 (11.22)
  Course 2: FU Week 24 (n=104) | 15.77 (11.17)
  Course 2: FU Month 9 (n=65) | 15.86 (11.67)
  Course 2: FU Month 12 (n=47) | 16.40 (10.68)
  Course 3: FU Week 8 (n=34) | 15.71 (11.44)
  Course 3: FU Week 16 (n=36) | 16.82 (12.53)
  Course 3: FU Week 24 (n=36) | 14.98 (11.21)
  Course 3: FU Month 9 (n=24) | 17.70 (12.49)
  Course 3: FU Month 12 (n=17) | 21.40 (12.74)

7. Secondary Outcome: Short-Form 36 (SF-36) Physical Composite Scores (PCS) by Treatment Course
Description: SF-36 was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the PCS and mental composite t-score (MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=171) | 34.57 (7.83)
  Course 1: FU Week 8 (n=165) | 36.28 (8.43)
  Course 1: FU Week 16 (n=160) | 37.23 (8.34)
  Course 1: FU Week 24 (n=161) | 37.94 (8.64)
  Course 1: FU Month 9 (n=74) | 37.28 (9.61)
  Course 1: FU Month 12 (n=39) | 36.92 (9.49)
  Course 2: FU Week 8 (n=102) | 37.27 (8.39)
  Course 2: FU Week 16 (n=105) | 38.34 (8.11)
  Course 2: FU Week 24 (n=103) | 39.17 (8.01)
  Course 2: FU Month 9 (n=66) | 38.68 (7.69)
  Course 2: FU Month 12 (n=48) | 37.34 (8.80)
  Course 3: FU Week 8 (n=33) | 37.95 (8.12)
  Course 3: FU Week 16 (n=35) | 39.43 (8.41)
  Course 3: FU Week 24 (n=36) | 37.62 (8.85)
  Course 3: FU Month 9 (n=23) | 37.99 (6.41)
  Course 3: FU Month 12 (n=15) | 34.95 (6.32)

8. Secondary Outcome: SF-36 MCS by Treatment Course
Description: SF-36 was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the PCS and MCS. The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=171) | 44.04 (12.76)
  Course 1: FU Week 8 (n=165) | 45.32 (12.42)
  Course 1: FU Week 16 (n=160) | 45.06 (12.06)
  Course 1: FU Week 24 (n=161) | 45.18 (12.59)
  Course 1: FU Month 9 (n=74) | 44.35 (13.38)
  Course 1: FU Month 12 (n=39) | 41.95 (14.30)
  Course 2: FU Week 8 (n=102) | 45.94 (11.34)
  Course 2: FU Week 16 (n=105) | 45.99 (11.71)
  Course 2: FU Week 24 (n=103) | 46.29 (11.89)
  Course 2: FU Month 9 (n=66) | 46.93 (13.56)
  Course 2: FU Month 12 (n=48) | 45.90 (12.33)
  Course 3: FU Week 8 (n=33) | 46.22 (10.79)
  Course 3: FU Week 16 (n=35) | 45.52 (13.41)
  Course 3: FU Week 24 (n=36) | 46.38 (12.20)
  Course 3: FU Month 9 (n=23) | 44.41 (13.96)
  Course 3: FU Month 12 (n=15) | 43.67 (13.73)

9. Secondary Outcome: SF-36 Domain Scores by Treatment Course - Physical Functioning
Description: as for outcome 8
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=172) | 43.26 (24.74)
  Course 1: FU Week 8 (n=170) | 46.80 (25.20)
  Course 1: FU Week 16 (n=164) | 46.85 (25.16)
  Course 1: FU Week 24 (n=164) | 49.58 (26.45)
  Course 1: FU Month 9 (n=76) | 47.30 (26.17)
  Course 1: Follow-up Month 12 (n=39) | 46.92 (30.21)
  Course 2: FU Week 8 (n=105) | 47.17 (24.51)
  Course 2: FU Week 16 (n=106) | 49.03 (24.91)
  Course 2: FU Week 24 (n=107) | 51.10 (24.23)
  Course 2: FU Month 9 (n=66) | 50.50 (22.87)
  Course 2: FU Month 12 (n=49) | 47.41 (23.62)
  Course 3: FU Week 8 (n=35) | 48.01 (26.63)
  Course 3: FU Week 16 (n=37) | 51.35 (26.84)
  Course 3: FU Week 24 (n=38) | 46.32 (28.44)
  Course 3: FU Month 9 (n=25) | 48.23 (26.16)
  Course 3: FU Month 12 (n=17) | 48.99 (29.37)

10. Secondary Outcome: SF-36 Domain Scores by Treatment Course - Bodily Pain
Description: as for outcome 8
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=172) | 37.22 (18.00)
  Course 1: FU Week 8 (n=169) | 46.06 (20.62)
  Course 1: FU Week 16 (n=164) | 47.98 (22.29)
  Course 1: FU Week 24 (n=164) | 48.70 (21.39)
  Course 1: FU Month 9 (n=75) | 46.55 (25.29)
  Course 1: FU Month 12 (n=39) | 44.10 (25.24)
  Course 2: FU Week 8 (n=105) | 47.15 (20.93)
  Course 2: FU Week 16 (n=106) | 50.34 (21.60)
  Course 2: FU Week 24 (n=104) | 51.38 (22.71)
  Course 2: FU Month 9 (n=66) | 51.23 (20.68)
  Course 2: FU Month 12 (n=48) | 48.58 (24.00)
  Course 3: FU Week 8 (n=35) | 47.60 (18.98)
  Course 3: FU Week 16 (n=36) | 51.94 (18.94)
  Course 3: FU Week 24 (n=38) | 47.92 (21.00)
  Course 3: FU Month 9 (n=25) | 43.24 (19.15)
  Course 3: FU Month 12 (n=16) | 32.56 (18.49)

11. Secondary Outcome: SF-36 Domain Scores by Treatment Course - Physical Role Functioning
Description: SF-36 was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the physical and mental composite t-scores (PCS and MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=173) | 45.85 (23.75)
  Course 1: FU Week 8 (n=170) | 50.04 (24.11)
  Course 1: FU Week 16 (n=166) | 51.28 (24.43)
  Course 1: FU Week 24 (n=165) | 52.92 (24.15)
  Course 1: FU Month 9 (n=76) | 49.51 (25.41)
  Course 1: FU Month 12 (n=39) | 47.44 (25.80)
  Course 2: FU Week 8 (n=103) | 52.79 (24.09)
  Course 2: FU Week 16 (n=106) | 53.54 (21.54)
  Course 2: FU Week 24 (n=107) | 55.32 (23.11)
  Course 2: FU Month 9 (n=66) | 56.91 (20.89)
  Course 2: FU Month 12 (n=49) | 52.98 (20.19)
  Course 3: FU Week 8 (n=35) | 52.32 (21.55)
  Course 3: FU Week 16 (n=36) | 53.47 (25.64)
  Course 3: FU Week 24 (n=38) | 50.99 (23.41)
  Course 3: FU Month 9 (n=24) | 51.82 (23.05)
  Course 3: FU Month 12 (n=17) | 44.49 (22.84)

12. Secondary Outcome: SF-36 Domain Scores by Treatment Course - Emotional Role Functioning
Description: SF-36was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the physical and mental composite t-scores (PCS and MCS). The range for all 8 domains as well as for the composite t-scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=173) | 57.80 (27.52)
  Course 1: FU Week 8 (n=170) | 61.91 (26.27)
  Course 1: FU Week 16 (n=166) | 60.44 (28.06)
  Course 1: FU Week 24 (n=165) | 62.12 (26.87)
  Course 1: FU Month 9 (n=76) | 56.52 (28.52)
  Course 1: FU Month 12 (n=39) | 55.98 (30.82)
  Course 2: FU Week 8 (n=104) | 61.30 (25.41)
  Course 2: FU Week 16 (n=106) | 62.74 (25.28)
  Course 2: FU Week 24 (n=107) | 61.53 (25.41)
  Course 2: FU Month 9 (n=66) | 62.75 (26.28)
  Course 2: FU Month 12 (n=49) | 61.05 (23.22)
  Course 3: FU Week 8 (n=34) | 60.29 (25.55)
  Course 3: FU Week 16 (n=37) | 61.26 (29.35)
  Course 3: FU Week 24 (n=38) | 60.53 (26.04)
  Course 3: FU Month 9 (n=24) | 54.51 (31.37)
  Course 3: FU Month 12 (n=17) | 55.39 (25.84)

13. Secondary Outcome: SF-36 Domain Scores by Treatment Course - Emotional Well-Being
Description: as for outcome 8
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=171) | 61.71 (21.25)
  Course 1: FU Week 8 (n=169) | 64.38 (20.36)
  Course 1: FU Week 16 (n=164) | 64.70 (20.02)
  Course 1: FU Week 24 (n=165) | 64.26 (20.77)
  Course 1: FU Month 9 (n=76) | 64.08 (23.23)
  Course 1: FU Month 12 (n=39) | 57.85 (24.50)
  Course 2: FU Week 8 (n=105) | 65.44 (19.45)
  Course 2: FU Week 16 (n=106) | 65.33 (19.75)
  Course 2: FU Week 24 (n=106) | 66.45 (19.63)
  Course 2: FU Month 9 (n=66) | 67.67 (20.60)
  Course 2: FU Month 12 (n=49) | 65.82 (19.75)
  Course 3: FU Week 8 (n=35) | 66.43 (18.01)
  Course 3: FU Week 16 (n=37) | 63.99 (24.25)
  Course 3: FU Week 24 (n=38) | 65.46 (20.87)
  Course 3: FU Month 9 (n=25) | 62.80 (20.82)
  Course 3: FU Month 12 (n=16) | 61.88 (21.20)

14. Secondary Outcome: SF-36 Domain Scores by Treatment Course - Social Functioning
Description: as for outcome 8
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=173) | 66.47 (25.39)
  Course 1: FU Week 8 (n=171) | 69.01 (26.55)
  Course 1: FU Week 16 (n=166) | 68.75 (25.63)
  Course 1: FU Week 24 (n=165) | 69.62 (26.77)
  Course 1: FU Month 9 (n=75) | 67.50 (27.34)
  Course 1: FU Month 12 (n=39) | 66.67 (30.26)
  Course 2: FU Week 8 (n=104) | 71.27 (24.44)
  Course 2: FU Week 16 (n=106) | 71.70 (24.60)
  Course 2: FU Week 24 (n=107) | 72.31 (25.76)
  Course 2: FU Month 9 (n=66) | 74.62 (27.21)
  Course 2: FU Month 12 (n=49) | 71.68 (24.84)
  Course 3: FU Week 8 (n=35) | 70.00 (23.13)
  Course 3: FU Week 16 (n=37) | 66.22 (25.15)
  Course 3: FU Week 24 (n=38) | 68.09 (24.95)
  Course 3: FU Month 9 (n=25) | 72.50 (24.74)
  Course 3: FU Month 12 (n=17) | 66.18 (32.71)

15. Secondary Outcome: SF-36 Domain Scores by Treatment Course - Vitality
Description: as for outcome 8
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=172) | 46.33 (20.61)
  Course 1: FU Week 8 (n=169) | 49.51 (21.04)
  Course 1: FU Week 16 (n=164) | 50.22 (20.86)
  Course 1: FU Week 24 (n=165) | 50.57 (21.99)
  Course 1: FU Month 9 (n=76) | 50.82 (22.53)
  Course 1: FU Month 12 (n=39) | 45.99 (22.77)
  Course 2: FU Week 8 (n=105) | 50.60 (20.59)
  Course 2: FU Week 16 (n=106) | 52.42 (20.94)
  Course 2: FU Week 24 (n=106) | 54.01 (21.81)
  Course 2: FU Month 9 (n=66) | 55.49 (19.19)
  Course 2: FU Month 12 (n=49) | 52.30 (18.47)
  Course 3: FU Week 8 (n=35) | 53.93 (24.12)
  Course 3: FU Week 16 (n=37) | 51.35 (24.57)
  Course 3: FU Week 24 (n=38) | 52.14 (24.33)
  Course 3: FU Month 9 (n=25) | 52.25 (26.01)
  Course 3: FU Month 12 (n=16) | 42.97 (23.92)

16. Secondary Outcome: SF-36 Domain Scores by Treatment Course - General Heath Perceptions
Description: as for outcome 8
Time Frame: Screening, FU Weeks 8, 16, and 24, and FU Months 9 and 12
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
scores on a scale
  Screening (n=173) | 45.74 (15.72)
  Course 1: FU Week 8 (n=171) | 47.46 (16.56)
  Course 1: FU Week 16 (n=166) | 50.82 (16.23)
  Course 1: FU Week 24 (n=164) | 50.65 (16.91)
  Course 1: FU Month 9 (n=76) | 49.38 (18.15)
  Course 1: FU Month 12 (n=39) | 46.15 (17.85)
  Course 2: FU Week 8 (n=104) | 50.32 (14.43)
  Course 2: FU Week 16 (n=106) | 52.04 (14.78)
  Course 2: FU Week 24 (n=107) | 52.93 (14.92)
  Course 2: FU Month 9 (n=66) | 51.04 (16.95)
  Course 2: FU Month 12 (n=49) | 48.98 (18.60)
  Course 3: FU Week 8 (n=35) | 52.27 (13.09)
  Course 3: FU Week 16 (n=37) | 52.14 (14.07)
  Course 3: FU Week 24 (n=37) | 52.90 (12.31)
  Course 3: FU Month 9 (n=25) | 50.54 (12.96)
  Course 3: FU Month 12 (n=17) | 45.29 (14.37)

17. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20 Percent (%), 50%, or 70% Improvement (ACR20/ACR50/ACR70) by Treatment Course
Description: ACR response was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). ACR20/50/70 response: ≥20/50/70%, respectively, improvement in SJC or TJC and 20/50/70% improvement in 3 of the following 5 criteria: 1) Physician's Global Assessment of Disease Activity, 2) Patient's Global Assessment of Disease Activity, 3) Patient's Assessment of Pain, 4) participants assessment of functional disability via HAQ-DI, and 5) C-reactive protein (CRP) or ESR at each visit.
Time Frame: 24 weeks after each course
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
percentage of participants
  Course 1: ACR20 (n=173) | 38.7
  Course 1: ACR50 (n=173) | 19.1
  Course 1: ACR70 (n=173) | 5.2
  Course 2: ACR20 (n=107) | 51.4
  Course 2: ACR50 (n=107) | 26.2
  Course 2: ACR70 (n=107) | 5.6
  Course 3: ACR20 (n=38) | 55.3
  Course 3: ACR50 (n=38) | 28.9
  Course 3: ACR70 (n=38) | 7.9

18. Secondary Outcome: Swollen Joint Count
Description: Mean sum of 28 swollen joints was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The 28 joints to be assessed for swelling were shoulder, elbow, wrist, metacarpophalangeal (MCP) joints 1-5, proximal interphalangeal (PIP) joints 1-5, and knee on both sides of the body. The sum of swollen joints ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status.
Time Frame: Screening and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
swollen joints
  Screening (n=165) | 8.52 (5.58)
  Course 1 FU Week 24 (n=165) | 4.09 (5.29)
  Course 2 FU Week 24 (n=105) | 3.65 (4.79)
  Course 3 FU Week 24 (n=37) | 3.51 (5.01)

19. Secondary Outcome: Tender Joint Count
Description: Mean sum of 28 tender joints was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). The 28 joints to be assessed for tenderness were shoulder, elbow, wrist, MCP joints 1-5, PIP joints 1-5, and knee on both sides of the body. The sum of tender joints ranged from 0 to 28 with 0 as best possible health status and 28 as worst health status.
Time Frame: Screening and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
tender joints
  Screening (n=165) | 12.92 (9.12)
  Course 1 FU Week 24 (n=165) | 7.32 (9.60)
  Course 2 FU Week 24 (n=105) | 6.31 (7.88)
  Course 3 FU Week 24 (n=37) | 7.00 (9.02)

20. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: Physician's Global Assessment of Disease Activity was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). Baseline was defined as the original baseline score from assessment performed in Study ML19070. Physicians were to assess the disease activity on a 100-mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right hand extreme (100 mm) as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: Baseline and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
mm
  Baseline (n=167) | 64.17 (15.12)
  Course 1 Week 24 (n=167) | 28.50 (22.23)
  Course 2 Week 24 (n=106) | 27.67 (24.32)
  Course 3 Week 24 (n=38) | 28.82 (22.52)

21. Secondary Outcome: Patient's Global Assessment of Disease Activity
Description: Patient Global Assessment of Disease Activity was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). Baseline was defined as the original baseline score from assessment performed in Study ML19070. Participants were to assess the disease activity on a 100-mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right hand extreme (100 mm) as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: Baseline and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
mm
  Baseline (n=164) | 63.40 (21.10)
  Course 1 Week 24 (n=164) | 34.13 (23.60)
  Course 2 Week 24 (n=107) | 34.50 (23.17)
  Course 3 Week 24 (n=38) | 33.66 (23.77)

22. Secondary Outcome: Patient's Assessment of Pain
Description: Patient Assessment of Pain was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). Baseline was defined as the original baseline score from assessment performed in Study ML19070. Participants were to assess their current level of pain on a 100 mm horizontal VAS. The left-hand extreme of the line (0 mm) was described as "no pain" and the right-hand (100 mm) as "unbearable pain".
Time Frame: Baseline and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
mm
  Baseline (n=164) | 61.90 (21.26)
  Course 1 Week 24 (n=164) | 35.02 (23.50)
  Course 2 Week 24 (n=107) | 35.12 (23.15)
  Course 3 Week 24 (n=38) | 34.82 (25.63)

23. Secondary Outcome: C-Reactive Protein
Description: CRP measured in milligrams per deciliter (mg/dL) was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). Baseline was defined as the original baseline score from assessment performed in Study ML19070.
Time Frame: Baseline and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
mg/dL
  Baseline (n=164) | 1.82 (2.41)
  Course 1 Week 24 (n=164) | 0.89 (1.35)
  Course 2 Week 24 (n=105) | 0.88 (1.16)
  Course 3 Week 24 (n=38) | 0.84 (0.96)

24. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: ESR mean scores measured in mm/hr at was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). Baseline was defined as the original baseline score from assessment performed in Study ML19070.
Time Frame: Baseline and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
mm/hr
  Baseline (n=166) | 31.30 (19.66)
  Course 1 Week 24 (n=166) | 19.87 (14.20)
  Course 2 Week 24 (n=107) | 19.45 (16.42)
  Course 3 Week 24 (n=38) | 18.74 (11.59)

25. Secondary Outcome: Rheumatoid Factor (RF)
Description: RF measured in international units per milliliter (IU/mL) was assessed during follow-up at the specified timepoints following each course of treatment (participants could have received up to 3 courses of treatment with rituximab). Baseline was defined as the original baseline score from assessment performed in Study ML19070.
Time Frame: Baseline and Week 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Rituximab Plus MTX
Number analyzed (Participants) | 173
IU/mL
  Baseline (n=158) | 187.18 (339.42)
  Course 1 Week 24 (n=158) | 70.16 (163.80)
  Course 2 Week 24 (n=102) | 63.17 (144.50)
  Course 3 Week 24 (n=38) | 58.52 (117.73)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Rituximab Plus MTX
Serious Adverse Events (participants affected / at risk) | 47/193
Other Adverse Events (participants affected / at risk) | 105/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus MTX (N=193)
Gangrene (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Hepatic enzyme increased (Investigations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Genital haemorrhage (Reproductive system and breast disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Coronary artery stenosis (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Toxic nodular goitre (Endocrine disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Chronic sinusitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus MTX (N=193)
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Dilatation ventricular (Cardiac disorders) | 1
Heart valve insufficiency (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Blindness transient (Eye disorders) | 1
Cataract (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 2
Erythema of eyelid (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 5
Glossitis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Reflux oesophagitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 5
Impaired healing (General disorders) | 1
Infusion related reaction (General disorders) | 7
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Allergy to arthropod sting (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Acute tonsillitis (Infections and infestations) | 3
Borrelia infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 17
Cystitis (Infections and infestations) | 3
Eye infection bacterial (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 8
Gastrointestinal infection (Infections and infestations) | 1
Herpes ophthalmic (Infections and infestations) | 2
Herpes simplex (Infections and infestations) | 2
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Hordeolum (Infections and infestations) | 1
Infected epidermal cyst (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Laryngitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 43
Onychomycosis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 5
Otitis media (Infections and infestations) | 2
Paronychia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 8
Rhinitis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 5
Tinea pedis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 4
Epicondylitis (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 2
Tendon rupture (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Body temperature increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Migraine (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 6
Depressive symptom (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Psychotic disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Transient psychosis (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 2
Menopausal symptoms (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Acrodermatitis (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Rash papular (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Urticaria localised (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 7
Hypertensive crisis (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Eyelid oedema (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.